CLINICAL TRIAL: NCT02152488
Title: Cerebral Blood Flow During Flexion and Rotation of the Cervical Spine
Acronym: TCDPOS
Status: Completed | Type: Observational
Sponsor: University Hospital Schleswig-Holstein (Other)
Responsible Party: Principal Investigator, Axel Fudickar, Dr. med., University Hospital Schleswig-Holstein
Other Study IDs: Fudickar4
Record Dates: First submitted 2014-05-21; First posted 2014-06-02 (Estimated); Last update posted 2014-06-02 (Estimated); Status verified 2014-05

CONDITIONS: Functional Blood Flow Disorder
Keywords: cerebral blood flow; position; cervical spine

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Rotation or flexion of the cervical spine is unavoidable during positioning for some surgical procedures as carotid endarterectomy, thyroidectomy and surgery of the shoulder. Rotation or flexion may reduce blood flow in the carotid or vertebral arteries and induce intraoperative cerebral ischemia with impact on the neurological outcome of surgery. Predominantly if the circulus willisii is incomplete because of congenital variation, collateral arteries may not be sufficient to compensate reduced blood flow in one carotid or vertebral artery. This may be aggravated by intraoperative hypotension in limits tolerable under normal conditions but fatal during impairment of vascular conductivity by positioning. The middle cerebral artery (MCA) is a final large scale pathway of cerebral blood flow and hence relevant reduction of flow in the MCA may serve as a surrogate parameter for relevant reduction of cerebral blood flow caused by carotid stretching or narrowing.

Objective of this study is to investigate, if MCA blood flow in normal male and female subjects, aged 18 to 85 years, is reduced in extended and rotated cervical spine position in comparison to neutral position.

DETAILED DESCRIPTION:
Blood flow in the middle cerebral artery (MCA) was measured bilaterally using a bidirectional multigate 2Mhz pulsed wave Transcranial Doppler (Multidop T1, Software Multiflow MF version 8.27j, DWL Corp., Sipplingen, Germany). Using a trans-temporal approach to the proximal segment (M1) of the MCA, the Doppler probes were fixed bilaterally with an adjustable mounting (SPENCER helmet) to keep the angle and depth of insonation constant over time. With the upper cervical spine in a neutral sagittal orientation, the insonation depth was chosen between 45 and 55 mm and the point permitting best recording was fixed. A sample volume of 5 mm, a sonographic frequency of 128 Hz FFT, and a fast sweep for temporal overlap were determined. Low power and low gain was set within the dynamic range of the system. All measurements were performed between 10:00 AM and 2:00 PM, by the same examiner (JL) in a quiet, warm, well-lit room. Each subject was asked to assume a relaxed, supine position. Patients eyes were closed to eliminate stimulation of the occipital cortex. Three minutes rest were provided to acclimatize and stabilize haemodynamically. Non-invasive blood pressure was measured at both arms before and after the procedure to ensure that any possible changes in blood flow were not related to blood pressure changes. The time-averaged mean blood flow velocities on both sides were measured with the cervical spine in neutral position, rotated maximally to the left, then to the right, hyperextended and then hyperextended and rotated to the left and to the right position. Measurements were performed after 1 min of stable blood flow. Neutral position was reestablished after each position and next maneuver started after blood velocities in neutral position had normalized to velocities in starting neutral position.

ELIGIBILITY:
Inclusion Criteria:

* Patients presenting ambulant for preoperative evaluation for routine surgery.

Exclusion Criteria:

* Cranial spine pathology and cerebral vascular disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 80 patients presenting in the pre-anaesthesia ambulance of the University Hospital Schleswig-Holstein, Campus Kiel were enrolled in the study. Exclusion criteria were cranial spine pathology and known cerebral vascular disease.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2010-03; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
Blood flow in middle cerebral artery during rotation of the cervical spine | From measurement of baseline blood flow until measurement of blood flow during rotation to the right and hyperextension of the cervical spine up to 1 hour
  Blood flow in the middle cerebral artery (MCA) was measured bilaterally using a bidirectional multigate 2Mhz pulsed wave Transcranial Doppler in normal and rotated position of the cervical spine.

CONTACTS AND LOCATIONS:
Overall Officials: Axel Fudickar, Dr., Principal Investigator — University Hospital Schleswig-Holstein
Locations (1):
- University Hospital Schleswig-Holstein, Campus Kiel, Kiel, Schleswig-Holstein, Germany